CLINICAL TRIAL: NCT03365297
Title: Targeted Drug Intervention to Inhibit Cancer Progression in Men on Active Surveillance for Prostate Cancer. Therapeutics in Active Prostate Cancer Surveillance (TAPS01)
Brief Title: Therapeutics in Active Prostate Cancer Surveillance
Acronym: TAPS01
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: CCTU- Cancer Theme (Other)
Collaborators: Janssen-Cilag Ltd. (Industry)
Responsible Party: Sponsor-Investigator, CCTU- Cancer Theme, CCTU Cancer Theme, Cambridge University Hospitals NHS Foundation Trust
Organization: Cambridge University Hospitals NHS Foundation Trust (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: TAPS01; 2017-001700-29 (EudraCT Number)
Record Dates: First submitted 2017-11-21; First posted 2017-12-07 (Actual); Last update posted 2019-11-19 (Actual); Status verified 2018-06

CONDITIONS: Prostate Cancer
MeSH Terms: conditions — Prostatic Neoplasms | interventions — apalutamide

STUDY DESIGN:
Intervention Model Description: Single centre, single arm open labelled Phase II window study
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Treatment (Experimental): apalutamide, 240mg (4x60mg tablets) orally, daily for a max. duration of 90 continuous days.
  Interventions: Drug: Apalutamide

INTERVENTIONS:
Drug: Apalutamide — 240mg (4x60mg) oral tablets daily over a max. of 90 days
  Other Names: ARN509; JNJ-56021927

SUMMARY:
Testing if short-term use of apalutamide can reduce image defined tumour volumes in men with detectable lesion on multi-parametric Magnetic Resonance Imaging (mpMRI) and being managed by Active Surveillance. The trial will also evaluate the tolerability and side effect profile of men on AS using short term apalutamide and patient acceptability as a therapeutic strategy, as well as determining feasibility of a larger prospective randomised trial of apalutamide.

DETAILED DESCRIPTION:
The numbers of men diagnosed with prostate cancer in the United Kingdom (UK) and worldwide is increasing. In the UK 46,690 men were diagnosed in 2014 alone and it is estimated this figure will be closer to 70,000 by 2030. A significant proportion of these men will present with organ confined and low or intermediate risk disease. There is increasing recognition that many men with low and intermediate risk prostate cancer do not need immediate radical therapy.

There is sufficient evidence that pharmacological intervention used as short-term therapy in men with low to intermediate-risk disease can inhibit the growth of prostate tumours and delay or remove the need for radical therapy in men managed by active surveillance. Given the irrefutable role of the androgen receptor in prostate cancer pathogenesis it is logical to target this pathway as a method of inhibiting or delaying disease progression.

This window study will be built on the known anti-androgen effects of apalutamide and investigate the efficacy of using it as a short intervention strategy to cause a physiological change in the tumour by reducing its volume. Tumour volume can be measured using the well-established place of mpMRI defined tumour volumes as a surrogate of disease presence and change. The rationale for a short duration treatment is that it will not have the long term debilitating effects of androgen deprivation on general health and prevent the onset of androgen resistance.

It is anticipated that if successful, this approach could be a new therapeutic strategy for these men who otherwise are living and waiting for their disease to progress or not.

ELIGIBILITY:
Inclusion Criteria:

* Given Informed Consent (IC) to participate
* Age 18 or over
* Eastern Cooperative Oncology Group (ECOG) status 0-2
* Diagnosed with prostate cancer
* Patient selection of active surveillance as a management option
* mpMRI detectable lesion
* Prostate cancer on biopsy from a mpMRI defined lesion
* No contraindications to apalutamide
* Normal full blood count and normal renal and liver function tests
* At least 6 months since initiation of active surveillance and/or last rebiopsy date.
* Low or intermediate risk prostate cancer according to National Institute for Health and Care Excellence (NICE) classification
* M score of ≥ 3 using Prostate Imaging Reporting and Data System (PIRADS) version 2 reporting criteria

Exclusion Criteria:

* Contraindications to apalutamide or its excipients
* Concurrent medication that can lower seizure threshold
* Prior localised therapy for prostate cancer
* Any prior use of androgen deprivation therapy or androgen receptor targeting agents
* Any prior systemic therapy for prostate cancer
* Patient unable to have prostate 3T mpMRI scan
* Presence of any pelvic or hip metalwork

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 11 (Actual)
Dates: Start 2018-06-05 (Actual); Primary Completion 2019-07-25 (Actual); Study Completion 2019-07-25 (Actual)

PRIMARY OUTCOMES:
Physiological Response | over a 90 day treatment period
  Tumour volume downsizing/absence of lesion, as determined by mpMRI

SECONDARY OUTCOMES:
Patient Reported Outcomes | over 120 days
  Function and wellbeing using established standardised EQ-5D-5L and EORTC-QLQ30+PR25 module questionnaires
Adverse Events | over 120 days
  tolerability and side effect profile

OTHER OUTCOMES:
Patient acceptability | over an estimated 1 year recruitment period
  number of men approached versus recruited

CONTACTS AND LOCATIONS:
Overall Officials: Vincent J Gnanapragasam, Principal Investigator — Cambridge University Hospitals NHS Foundation Trust/University of Cambridge
Locations (1):
- Cambridge University Hospitals NHS Foundation Trust/Addenbrookes Hospital, Cambridge, Cambridgeshire, United Kingdom

IPD SHARING:
Plan to Share IPD: No